CLINICAL TRIAL: NCT03232034
Title: The Role of Dietary Milk Minerals and Protein in Gut Hormone Secretion
Brief Title: Calcium, Protein and Gut Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Lecturer (Assistant Professor) in Human Physiology, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: REACH EP 16/17_164
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Diabetes
Keywords: Calcium citrate, dairy product, whey protein, appetite, metabolism
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Calcium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and Researchers will be blinded to the interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Calcium Citrate (Placebo Comparator): Calcium citrate (1000 mg calcium) will be consumed by participants in the morning between 8-10 am after 8-14 h fasting. Blood samples, appetite scales and expired breath samples will be taken in a regular intervals for 2 h after ingestion.
  Interventions: Dietary Supplement: Calcium Citrate
- Milk Mineral Supplement (Active Comparator): Milk mineral supplement (equating to 1000 mg calcium) will be consumed by participants in the morning between 8-10 am after 8-14 h fasting. Blood samples, appetite scales and expired breath samples will be taken in a regular intervals for 2 h after ingestion.
  Interventions: Dietary Supplement: Milk Mineral Supplement
- Milk mineral supplement plus Whey Protein Hydrolysate (Experimental): Milk mineral supplement (equating to 1000 mg calcium) plus whey protein hydrolysate (50 g) will be consumed by participants in the morning between 8-10 am after 8-14 h fasting. Blood samples, appetite scales and expired breath samples will be taken in a regular intervals for 2 h after ingestion.
  Interventions: Dietary Supplement: Milk Mineral Supplement; Dietary Supplement: Whey Protein Hydrolysate

INTERVENTIONS:
Dietary Supplement: Calcium Citrate — 1000 mg calcium as calcium citrate
  Arms: Calcium Citrate
Dietary Supplement: Milk Mineral Supplement — Milk Minerals containing 1000 mg calcium
  Arms: Milk Mineral Supplement; Milk mineral supplement plus Whey Protein Hydrolysate
Dietary Supplement: Whey Protein Hydrolysate — 50 g whey protein hydrolysate
  Arms: Milk mineral supplement plus Whey Protein Hydrolysate

SUMMARY:
Gut hormones have therapeutic potential in the prevention and treatment obesity and type 2 diabetes (T2D). Milk protein and calcium can each potentiate gut hormones following meal ingestion in humans. However, these nutrients may interact synergistically (and with other minerals in milk) such that specific co-ingestion of these nutrients is required to obtain the full therapeutic potential for metabolism and energy balance. This proposal is to perform a pilot study on the effect of co-ingesting Capolac® plus protein on circulating gut hormone responses.

DETAILED DESCRIPTION:
Participants will be asked to arrive to the laboratory between 08:00 and 10:00 am after not eating for between 8-14 hours i.e. in a fasted state (water intake is permitted and encouraged). Participants will then be given one of three test drinks: 1) calcium citrate (1000 mg); 2) milk mineral supplement (equating to 1000 mg calcium); or 3) milk mineral supplement (equating to 1000 mg calcium) plus whey protein hydrolysate (50 g). Each of these drinks will also contain 500 mL of water and artificial sweetener (80 mg sucralose).

Blood samples will be taken before, and at 15, 30, 45, 60, 90 and 120 minutes after ingestion of the test drink to determine the concentrations of gut hormones (GIP, GLP-1 and PYY) circulating in the bloodstream. We will also ask participants to complete an appetite questionnaire at baseline and every 30 minutes after ingestion of the test drink to assess their appetite sensations. After the 120-minute time point, we will remove the cannula and the trial day will be complete.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women age between 18-65 yrs.
* Able to consume provided supplement.
* Weigh stable for the past 3 month (no change within 3%).

Exclusion Criteria:

* Any previous or current metabolic, cardio-pulmonary or musculoskeletal disease
* Not between the ages of 18-65 years
* A body mass index below 18.5 kg/m2 or above 30 kg/m2 (body mass (kg) divided by your height (m) squared)
* Taking medications that may influence your metabolism
* Plans to change your lifestyle (diet and/or physical activity) during the study period
* Not willing to refrain from alcohol containing drinks or unaccustomed exercise one day before the laboratory sessions.
* Current smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Postprandial plasma GLP-1 area under the curve (mmol/L x 120 min). | 120 min
  Plasma glucagon-like peptide-1 (GLP-1) concentrations

SECONDARY OUTCOMES:
Postprandial plasma GIP area under the curve (mmol/L x 120 min) | 120 min
  Plasma glucose-dependent insulinotropic peptide (GIP) concentrations
Postprandial plasma PYY area under the curve (mmol/L x 120 min) | 120 min
  Plasma peptide tyrosine tyrosine (PYY) concentrations.
Subjective ratings of appetite (au) | 120 min
  Visual analogue scales of appetite ratings
Energy metabolism (carbohydrate and fat oxidation) | 120 min
  Carbohydrate and fat oxidation (g/h) measured via indirect calorimetry
Postprandial plasma glucose | 120 min
  Plasma glucose concentrations (mmol/L).
Blood pressure | 120 min
  Systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

REFERENCES:
- [Derived] Chen YC, Smith HA, Hengist A, Chrzanowski-Smith OJ, Mikkelsen UR, Carroll HA, Betts JA, Thompson D, Saunders J, Gonzalez JT. Co-ingestion of whey protein hydrolysate with milk minerals rich in calcium potently stimulates glucagon-like peptide-1 secretion: an RCT in healthy adults. Eur J Nutr. 2020 Sep;59(6):2449-2462. doi: 10.1007/s00394-019-02092-4. Epub 2019 Sep 17. PMID 31531707